CLINICAL TRIAL: NCT03579615
Title: An Open-label, Single-centre, Randomised, Two-period, Cross-over Study to Assess the Efficacy and Safety of Day and Night Automated Closed-loop Glucose Control for 24 Hours in Adults With Type 1 Diabetes Comparing Faster-acting Insulin Aspart With Insulin Aspart
Brief Title: Comparison of Day and Night Closed-loop With Faster-acting Insulin Aspart With Insulin Aspart
Acronym: AP-MFT-01
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Manchester University NHS Foundation Trust (Other Government)
Collaborators: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: R04695
Record Dates: First submitted 2018-06-25; First posted 2018-07-06 (Actual); Last update posted 2022-08-22 (Actual); Status verified 2022-08

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Intervention Model Description: An open-label, single-centre, randomised, two-period, cross-over study
Masking Description: FIASP vs standard of care insulin
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- FIASP + closed loop device (Experimental): Subjects randomised to FIASP and closed loop device will be invited to have blood samples taken at baseline, CGM training, competency assessment, and optimisation of treatment. This is followed by inpatient stay where patients will be using FIASP + closed loop intervention for 24 hours. Participants will be advised to change their usual insulin to the corresponding study visit insulin formulation, 24 hours prior to admission. (For example; if the participant is on insulin aspart, this will be changed to faster-acting aspart 24-hour prior to the admission for closed loop with faster-acting aspart and vice versa).
  Interventions: Device: FIASP + closed loop device
- Insulin aspart (standard of care insulin) + closed loop device (Active Comparator): Subjects randomised to insulin aspart (standard of care insulin) and closed loop device will be invited to have blood samples taken at baseline, CGM training, competency assessment, and optimisation of treatment. This is followed by inpatient stay where patients will be using insulin aspart (standard of care insulin) + closed loop intervention for 24 hours.Participants will be advised to change their usual insulin to the corresponding study visit insulin formulation, 24 hours prior to admission. (For example; if the participant is on insulin aspart, this will be changed to faster-acting aspart 24-hour prior to the admission for closed loop with faster-acting aspart and vice versa).
  Interventions: Device: Insulin aspart (standard of care insulin) + closed loop device

INTERVENTIONS:
Device: FIASP + closed loop device — Participants will be advised to change their usual insulin to the corresponding study visit insulin formulation, 24 hours prior to admission. (For example; if the participant is on insulin aspart, this will be changed to faster-acting aspart 24-hour prior to the admission for closed loop with faster-acting aspart and vice versa).
  Arms: FIASP + closed loop device
Device: Insulin aspart (standard of care insulin) + closed loop device — Participants will be advised to maintain their usual insulin 24 hours prior to admission.
  Arms: Insulin aspart (standard of care insulin) + closed loop device

SUMMARY:
The main objective of the study is to determine whether automated closed-loop using faster-acting insulin aspart will improve glucose control and reduce the burden of hypoglycaemia over a 23-hour period compared to insulin aspart under conditions mimicking under-estimation of meal carbohydrate content or missed meal bolus. Faster-acting insulin aspart (FIASP) is a novel formulation of insulin aspart in which two additional excipients (L-arginine and Niacinamide) have been added, resulting in accelerated initial absorption and more than double the glucose lowering effect in the first 30 minutes after subcutaneous administration using insulin pump. To date, no closed-loop study has been performed to evaluate the benefit of faster-acting aspart over insulin aspart during closed-loop system use.

DETAILED DESCRIPTION:
This is an open-label, single-centre, two-period, randomised, cross over study. The study involves a screening visit to assess participant eligibility and two 24 hour in-patient stays at the clinical research facility during which day and night glucose levels will be controlled by the closed-loop system with either faster-acting insulin aspart or insulin aspart.

Up to 22 adults with type 1 diabetes and treated with continuous subcutaneous insulin infusion will be recruited, aiming for 16 completed participants. Recruitment will take place at Manchester Diabetes Centre, Manchester Royal Infirmary, Manchester, UK. Participants will attend the Manchester Clinical Research Facility (MCRF), Manchester, on two occasions. In random order, they will undergo two closed-loop study days using either faster-acting insulin aspart or insulin aspart. During the study days, the closed-loop control algorithm will automatically modulate d insulin infusion rate based on real-time subcutaneous glucose sensor measurements. Participants will receive standardised meals with half usual meal bolus for the evening meal and no meal bolus for lunch time meal during each study day.

ELIGIBILITY:
Inclusion Criteria:

1. The subject is 18 years and older
2. The subject has type 1 diabetes, as defined by WHO for at least 1 year or is confirmed C-peptide negative
3. The subject will have been an insulin pump user for at least 3 months
4. The subject is treated with any of the rapid acting insulin analogues
5. The subject is willing to adhere to study procedures
6. HbA1c ≥ 7.0% (53 mmol/mol) and ≤ 10 % (86mmol/mol) based on analysis from local laboratory or equivalent within 3 months prior to enrolment
7. The subject is literate in English

Exclusion Criteria:

* 1. Non-type 1 diabetes mellitus including those secondary to chronic disease 2. Any other physical or psychological disease likely to interfere with the normal conduct of the study 3. Untreated celiac disease or hypothyroidism 4. Current treatment with drugs known to interfere with glucose metabolism, e.g. systemic corticosteroids, Metformin, SGLT2 inhibitors, non-selective beta-blockers and MAO inhibitors etc.

  5. Known or suspected allergy against insulin 6. Subjects with clinical significant nephropathy, neuropathy or proliferative retinopathy as judged by the investigator 7. Total daily insulin dose > 2 U/kg/day 8. Total daily insulin dose < 10 U/day 9. Pregnancy, planned pregnancy, or breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2020-12-23 (Actual); Primary Completion 2022-02-24 (Actual); Study Completion 2022-08-01 (Actual)

PRIMARY OUTCOMES:
Time spent in the target glucose range | 23 hours
  Time spent in the target glucose range between 3.9 to 10.0 mmol/l (70 to 180mg/dl) based on sensor glucose levels between the hours of 19:00 on day 1 and 18:00 hours on day 2 of the inpatient stay.

SECONDARY OUTCOMES:
Time spent in the target glucose range within 4 hours of each meal | 4 hours
  Time spent in the target glucose range between 3.9 to 10.0 mmol/l (70 to 180mg/dl) based on sensor glucose levels during the first 4 hours following each meal
Incremental area under the curve of sensor glucose level within 4 hours of each meal | 4 hours
  Incremental area under the curve of sensor glucose level during the first 4 hours after each meal
Time spent below target glucose | 23 hours
  Time spent below target glucose (<3.9mmol/l) (<70mg/dl)
Time spent above target glucose | 23 hours
  Time spent above target glucose (10.0 mmol/l) (180 mg/dl)
Average, coefficient of variation and standard deviation glucose levels | 23 hours
  Average, coefficient of variation and standard deviation glucose levels
The time with sensor glucose levels < 3.5 mmol/l (63 mg/dl) | 23 hours
  The time with sensor glucose levels < 3.5 mmol/l (63 mg/dl)
The time with sensor glucose levels <3.0 (54mg/dl) | 23 hours
  The time with sensor glucose levels <3.0 (54mg/dl)
The time with sensor glucose levels <2.8 mmol/l (50 mg/dl) | 23 hours
  The time with sensor glucose levels <2.8 mmol/l (50 mg/dl)
The time with sensor glucose levels in the significant hyperglycaemia | 23 hours
  The time with sensor glucose levels in the significant hyperglycaemia (glucose levels > 16.7 mmol/l) (300mg/dl)
Total, basal and bolus insulin dose | 23 hours
  Total, basal and bolus insulin dose
AUC of glucose below 3.0mmol/l (54mg/dl) | 23 hours
  AUC of glucose below 3.0mmol/l (54mg/dl)

CONTACTS AND LOCATIONS:
Locations (1):
- Manchester University Hospitals NHS Foundation Trust, Manchester, United Kingdom

REFERENCES:
- [Derived] Thabit H, Mubita W, Rubio J, Karuppan M, Schofield J, Willinska ME, Hovorka R, Leelarathna L. Comparison of faster-acting aspart with insulin aspart under conditions mimicking underestimation or missed meal boluses in type 1 diabetes using closed-loop insulin delivery. Diabetes Obes Metab. 2023 Apr;25(4):1121-1124. doi: 10.1111/dom.14942. Epub 2022 Dec 27. No abstract available. PMID 36514847